CLINICAL TRIAL: NCT03284749
Title: Randomised Controlled Trial on the Effect of Copper Impregnated Dressings and Maternity Pads on the Healing of Obstetric Wounds and Wound Infection
Brief Title: Effect of Copper on the Healing of Obstetric Wounds
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croydon Health Services NHS Trust (Other)
Responsible Party: Principal Investigator, Mr Abdul H Sultan, Consultant Obstetrician and Gynaecologist, Croydon Health Services NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15/07
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Cesarean Section; Infection; Perineal Infection; Wound Infection; Surgical Site Infection
Keywords: Copper Oxide; Antibiotic Resistance
MeSH Terms: conditions — Infections; Wound Infection; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: All women are randomised to either the copper or the control group. Randomisation will be done separately for the caesarean section and vaginal delivery group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After inclusion all patients will be randomised for a wound dressing or maternity pad with (study group) or without copper (control group). The two sets of wound dressings and pads will be marked "A" or "B". Both the clinician and the patient will be blinded to the randomised group. Only the manufacturer will be aware of which group contains copper.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Copper impregnated wound dressing (Experimental): Wound dressing impregnated with 3% copper oxide ions, to be applied for 7 days after caesarean section
  Interventions: Other: Copper impregnated wound dressing
- Normal wound dressing (Placebo Comparator): Wound dressing without copper, to be applied for 7 days after caesarean section
  Interventions: Other: Normal wound dressing
- Copper impregnated maternity pads (Experimental): Maternity pads impregnated with 3% copper oxide ions, to be used for 14 days after delivery
  Interventions: Other: Copper impregnated maternity pads
- Normal maternity pads (Placebo Comparator): Maternity pads without copper, to be used for 14 days after delivery
  Interventions: Other: Normal maternity pads

INTERVENTIONS:
Other: Copper impregnated wound dressing — Copper impregnated wound dressing
  Arms: Copper impregnated wound dressing
Other: Normal wound dressing — Normal wound dressing
  Arms: Normal wound dressing
Other: Copper impregnated maternity pads — Copper impregnated maternity pads
  Arms: Copper impregnated maternity pads
Other: Normal maternity pads — Normal maternity pads
  Arms: Normal maternity pads

SUMMARY:
The most common complication of vaginal delivery is perineal tearing with a prevalence of 85% and 70% will need suturing. The caesarean section rate worldwide is rising and the rate in Croydon University Hospital is in the region of 25% of all deliveries. One in ten women will develop a wound infection of their perineal tear or caesarean section wound. Wound infection can cause pain, dehiscence, delayed wound healing, prolonged hospital stay, readmissions and interfere with a woman's ability to nurture their baby and enjoy motherhood. Copper has shown to have strong antimicrobial properties, with the ability to kill various bacteria including MRSA. It has also been shown that copper promotes new blood vessel formation and therefore enhance wound healing. This study is to investigate the effect of copper impregnated dressings and maternity pads on wound infection. Women will be randomised for a wound dressing or maternity pad with (study group) or without copper (control group). Both the clinician and the woman will be blinded to the randomised group. Wound infection will be assessed via a telephone questionnaire after 7, 14 and 30 days after delivery. When wound infection is suspected, based on the questionnaire, a swab of the wound site will be taken to detect the causative bacteria.

DETAILED DESCRIPTION:
This is a double blind randomised controlled pilot study to assess feasibility of copper impregnated wound dressings and maternity pads for the healing of obstetric wounds. All women having a caesarean section or with perineal sutures after a vaginal delivery will be recruited from the antenatal clinic (in case of an elective caesarean section) or from the maternity wards within Croydon Health Services. All women will be given a patient information sheet describing the study prior to consent and will be giving adequate time to read the information before signing the Informed consent. Participants will be followed up via a telephone questionnaire 7, 14 and 30 days after the delivery.

Randomisation:

After inclusion all participants will be randomised for a wound dressing or maternity pad with (study group) or without copper (control group). The two sets of wound dressings and pads will be marked "A" or "B". Both the clinician and the participant will be blinded to the randomised group. Only the manufacturer will be aware of which group contains copper.

Copper impregnated dressings:

As soon as possible, but within 12 hours after primary closure of the caesarean section incision, the randomised study dressing will be applied. The two study dressings were equivalent to the dressing normally used within this Trust, except the foam of one set of dressings was impregnated with 3% copper oxide ions. The two sets of wound dressings were marked "A" and "B" and both the women and clinician were blinded to the randomised group. According to local protocol the wound dressing will be left intact for 7 days following surgery and will be renewed if necessary.

Copper impregnated maternity pads As soon as possible, but within 12 hours after suturing, women will be asked to wear the study maternity pads, which will be provided. The two sets of study maternity pads will be equivalent to the currently recommended pads, except that one set of pads will have a thin top layer of non-woven polyester fibres with 3% copper oxide ions permanently attached to it. Women will be asked to use the pads for 14 days.

Patient data, history and physical examination:

Demographic data such as age, ethnicity, height and weight will be collected as well as obstetric data and delivery details. Past medical history such as concomitant (chronic) diseases and the use of medications will be obtained. Wound infection will be assessed via a telephone questionnaire after 7, 14 and 30 days after delivery. The data will be stored in a secure room within Trust facilities. All electronic data will be stored within password protected IT system within the Trust, which is only accessible by the clinical and research team.

Questionnaire:

For the assessment of surgical site infection, the Post Discharge Questionnaire used by the HPC surgical site infection surveillance will be used, which is according to the worldwide used definition of surgical site infection by the CDC.

Statistical analysis Statistical analysis will be performed using SPSS version 20.0 or higher. Infection rates in the perineal tear group and the caesarean section group will be analysed seperately. The infection rates in the study group (with copper) will be compared to the control group and possible risk factors for infection will be explored. the Chi-Square will be used to analyse categorical variables and the T-test or Mann Whitney-U test will be used to analyse continuous variables. Multivariable logistic regression will be used to investigate risk factors for development of infection.

Sample size calculation Since the effect of copper on infection rates is currently unknown, we will conduct a pilot study for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Delivered by caesarean section (emergency or elective), or vaginally, sustaining a perineal tear or episiotomy which needed to be sutured
* Ability to understand and read the content of the patient information sheet (in English, via an interpreter if needed and possible)
* Ability to give informed consent

Exclusion Criteria:

* Inability to give consent
* Fetal or neonatal death or poor neonatal outcome
* Obstetric anal sphincter injuries
* Included in another study on postpartum infection
* Wilson's disease
* Allergy to copper

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 774 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Post Discharge Questionnaire (PDQ) | 30 days
  Questionnaire used by the HPC for surgical site infection surveillance. Using worldwide definition of surgical site infection by the CDC infection is present if one of the 6 criteria are met: 1) discharge pus AND antibiotics prescribed; 2) Clinical signs* AND wound dehiscence; 3) Clinical signs* AND antibiotics prescribed; 4)Uterine tenderness AND antibiotics prescribed; 5) Abdominal tenderness AND antibiotics prescribed; 6) Purulent discharge from uterus AND antibiotics prescribed.
  * Clinical signs: at least 2 of pain, heat, redness or swelling

SECONDARY OUTCOMES:
Length of hospitalisation | 30 days
  Length of in hospital stay following child birth
Pain score | 7, 14 and 30 days after delivery
  Visual Analog Scale for wound pain

CONTACTS AND LOCATIONS:
Overall Officials: Abdul H Sultan, Principal Investigator — Croydon Health Services NHS Trust
Locations (1):
- Croydon Health Services NHS Trust, Croydon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson A, Thakar R, Sultan AH. Obstetric perineal wound infection: is there underreporting? Br J Nurs. 2012 Mar 8-21;21(5):S28, S30, S32-5. doi: 10.12968/bjon.2012.21.Sup5.S28. PMID 22489339
- [Background] American College of Obstetrics and Gynecology.. Operative vaginal delivery. Clinical management guidelines for obstetrician-gynecologists. American College of Obstetrics and Gynecology. Int J Gynaecol Obstet. 2001 Jul;74(1):69-76. doi: 10.1016/s0020-7292(01)00434-9. No abstract available. PMID 11480404
- [Background] Callwood A, Thomas J. The National Sentinel Caesarean Section Audit. Pract Midwife. 2000 Jun;3(6):34-5. No abstract available. PMID 11260996
- [Background] Smaill FM, Grivell RM. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. Cochrane Database Syst Rev. 2014 Oct 28;2014(10):CD007482. doi: 10.1002/14651858.CD007482.pub3. PMID 25350672
- [Background] Declercq E, Barger M, Cabral HJ, Evans SR, Kotelchuck M, Simon C, Weiss J, Heffner LJ. Maternal outcomes associated with planned primary cesarean births compared with planned vaginal births. Obstet Gynecol. 2007 Mar;109(3):669-77. doi: 10.1097/01.AOG.0000255668.20639.40. PMID 17329519
- [Background] Hillan EM. Postoperative morbidity following Caesarean delivery. J Adv Nurs. 1995 Dec;22(6):1035-42. doi: 10.1111/j.1365-2648.1995.tb03102.x. PMID 8675855
- [Background] Henderson E, Love EJ. Incidence of hospital-acquired infections associated with caesarean section. J Hosp Infect. 1995 Apr;29(4):245-55. doi: 10.1016/0195-6701(95)90271-6. PMID 7658004
- [Background] Ward VP, Charlett A, Fagan J, Crawshaw SC. Enhanced surgical site infection surveillance following caesarean section: experience of a multicentre collaborative post-discharge system. J Hosp Infect. 2008 Oct;70(2):166-73. doi: 10.1016/j.jhin.2008.06.002. Epub 2008 Aug 23. PMID 18723248
- [Background] Creech CB, Litzner B, Talbot TR, Schaffner W. Frequency of detection of methicillin-resistant Staphylococcus aureus from rectovaginal swabs in pregnant women. Am J Infect Control. 2010 Feb;38(1):72-4. doi: 10.1016/j.ajic.2009.06.015. Epub 2009 Oct 21. PMID 19836855
- [Background] ACOG Practice Bulletin No. 120: Use of prophylactic antibiotics in labor and delivery. Obstet Gynecol. 2011 Jun;117(6):1472-1483. doi: 10.1097/AOG.0b013e3182238c31. No abstract available. PMID 21606770
- [Background] Borkow G, Gabbay J. Copper as a biocidal tool. Curr Med Chem. 2005;12(18):2163-75. doi: 10.2174/0929867054637617. PMID 16101497
- [Background] Noyce JO, Michels H, Keevil CW. Potential use of copper surfaces to reduce survival of epidemic meticillin-resistant Staphylococcus aureus in the healthcare environment. J Hosp Infect. 2006 Jul;63(3):289-97. doi: 10.1016/j.jhin.2005.12.008. Epub 2006 May 2. PMID 16650507
- [Background] O'Gorman J, Humphreys H. Application of copper to prevent and control infection. Where are we now? J Hosp Infect. 2012 Aug;81(4):217-23. doi: 10.1016/j.jhin.2012.05.009. Epub 2012 Jun 26. PMID 22738611
- [Background] Borkow G, Gabbay J, Zatcoff RC. Could chronic wounds not heal due to too low local copper levels? Med Hypotheses. 2008;70(3):610-3. doi: 10.1016/j.mehy.2007.06.006. Epub 2007 Aug 6. PMID 17689198
- [Background] Sen CK, Khanna S, Venojarvi M, Trikha P, Ellison EC, Hunt TK, Roy S. Copper-induced vascular endothelial growth factor expression and wound healing. Am J Physiol Heart Circ Physiol. 2002 May;282(5):H1821-7. doi: 10.1152/ajpheart.01015.2001. PMID 11959648
- [Background] Uauy R, Olivares M, Gonzalez M. Essentiality of copper in humans. Am J Clin Nutr. 1998 May;67(5 Suppl):952S-959S. doi: 10.1093/ajcn/67.5.952S. PMID 9587135
- [Background] Hostynek JJ, Dreher F, Maibach HI. Human skin penetration of a copper tripeptide in vitro as a function of skin layer. Inflamm Res. 2011 Jan;60(1):79-86. doi: 10.1007/s00011-010-0238-9. Epub 2010 Aug 20. PMID 20721598

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03284749/Prot_SAP_000.pdf
  • Informed Consent Form (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT03284749/ICF_001.pdf